CLINICAL TRIAL: NCT00505869
Title: A Mood Management Intervention for Pregnant Smokers
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2004-0022
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Pregnancy; Smoking
Keywords: Pregnant Smokers; Mood Management Intervention; Health & Wellness Intervention; Smoking Cessation; Questionnaire; Survey
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Health; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva sample for cotinine.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Health & Wellness Intervention + Questionnaire
  Interventions: Behavioral: Health & Wellness Intervention; Behavioral: Questionnaire
- 2: Mood Management Intervention + Questionnaire
  Interventions: Behavioral: Questionnaire; Behavioral: Mood Management Intervention

INTERVENTIONS:
Behavioral: Health & Wellness Intervention — Counseling focusing on health concerns related to pregnancy, information about smoking and pregnancy, tips for quitting, and problem-solving skills to manage situations that might be triggers for smoking.
  Groups: 1
Behavioral: Questionnaire — Questionnaires about mood, confidence in quitting, smoking behavior, and social support.
  Other Names: Survey
Behavioral: Mood Management Intervention — Counseling focusing on learning to manage negative moods (depressed mood, tension, anxiety), as well as providing tips for quitting smoking, problem-solving skills, and information about smoking and pregnancy.
  Groups: 2

SUMMARY:
This proposal is aimed at testing the following hypotheses:

1. Cessation rates will be significantly greater for smokers in a mood management condition versus a health & wellness condition during pregnancy and at 3 and 6 months postpartum.
2. Pregnant smokers who have a higher level of depressive symptomatology will quit significantly less often in the health & wellness condition vs. mood management condition; those with a lower level of depressive symptomatology will not demonstrate this treatment difference.
3. Pregnant smokers who show higher levels of current depression at the start of the intervention will quit significantly less often than those smokers with lower levels.

The mood management intervention will result in higher levels of adaptive coping behavior, self-efficacy, social support, and perceived support from the counselor, and lower levels of negative affect, rumination, and perceived stress, than the health & wellness intervention and these variables will be related to abstinence. Thus, we will evaluate the effects of the intervention (health & wellness and mood management) on hypothesized treatment mechanisms, and assess the impact of those mechanisms on abstinence.

DETAILED DESCRIPTION:
Before treatment begins, you will have a screening visit with the study doctor/staff, to find out if you are eligible to take part in the study. This visit will involve an in-depth interview about your history of depression and other mental health problems. If you have not yet been to a doctor, the study staff will give you a urine pregnancy test to make sure you are pregnant.You will also be asked to complete several questionnaires regarding smoking history and other areas of your daily life. The questionnaires themselves take about 30-45 minutes to complete. The visit may last between 1 1/2 and 3 1/2 hours, depending on the complexity of the interview.

If you are eligible to take part in the study, you will receive one of two types of smoking cessation counseling. In one, counseling will focus on health concerns related to pregnancy, information about smoking and pregnancy, tips for quitting, and problem-solving skills to manage situations that might be triggers for smoking. In the other, counseling will focus on the learning to manage negative moods (depressed mood, tension, anxiety), as well as providing tips for quitting smoking, problem-solving skills, and information about smoking and pregnancy. Counseling sessions for both groups will last about an hour each.

During the first counseling visit, you will set a quit date for stopping smoking.

At each of the counseling visits, you will also be asked to provide a carbon monoxide (CO) measurement. This is done by blowing into a cardboard tube attached to a CO monitor. This will show whether or not you are still smoking. You will also complete several questionnaires at every visit, which will take about 20-40 minutes. These questionnaires will include questions about your mood, confidence in quitting, smoking behavior, and social support.

Four times during the study, you will provide a saliva sample for tests to look for cotinine, a chemical produced by the breakdown of nicotine during smoking. This sample will be taken using a dental roll (cotton swab) placed in the mouth for several minutes to absorb saliva. Like the CO test, this test will help researchers measure how much you are smoking.

You will be asked to attend a maximum of 12 individual counseling sessions, over a 2-3 month period. Also, you will receive 4 follow-up telephone calls from the study staff. These calls will take place 2 weeks after treatment ends, 2 weeks before your due date, 2 weeks after your delivery, and 4 weeks after your delivery.

Additional in-person clinic visits will take place at 3- and 6-months after your delivery. During these visits you will be asked to provide carbon monoxide (CO) and cotinine measurements of your smoking and to complete a packet of questionnaires regarding your mood, social support, and smoking behavior.

So that the study researchers can keep in contact with you throughout the study and over the long period of time between your end of treatment visit and the 3- and 6-month postpartum follow-up visits, you will be asked at the baseline visit to provide the name and address of 3 contacts (family members/friends) that you feel confident would have updated contact information on you. You will also be asked to sign a letter giving your contacts permission to provide your updated information to the study staff. The staff will check this contact information at the end-of-treatment visit, at one of the telephone assessment calls and then again at the 3-month follow-up visit.

If the study staff is not able to reach you by phone, mail, or the information provided by your contacts, they may attempt to locate you through telephone directory assistance (411) or internet search sources (for example, Google or Yahoo!), which use information from the public domain (meaning everyone has access to it).

If the study staff is still unable to locate your new contact information, they may use a locator service such as Transunion or the National Change of Address (NCOA) database maintained by the United States Postal Service, as a last resort. Transunion uses things like magazine subscriptions and credit applications to find new addresses, and the NCOA uses the Change of Address cards filed with the post office when a person moves and requests their mail be forwarded to a new address. If the study staff has to use either of these services, they would only disclose your name and last known address.

Researchers may also use Temporary Assistance for Needy Families (Welfare)/Medicaid Administrative databases, maintained by the Texas Department of Human Services (TDHS), to find contact information for participants who cannot be found for follow-up study. The study staff will provide designated Welfare personnel with a list containing the name, date of birth, last known address, and other relevant personal identifiers for each of the participants with whom we cannot contact. In return, Welfare personnel will provide study staff with the most recent locator information (such as address and phone numbers) for each of the listed participants.

Under certain circumstances, your counselor may provide counseling to you over the phone. Additionally, you may be mailed some questionnaires and/or a cotinine sample kit. If so, a pre-addressed, postage paid envelope will be provided for the return of these materials.

Each of the counseling sessions will be videotaped. In addition, the SCID assessment done at the Baseline visit and the LIFE Assessment done at both follow-up visits, may be videotaped or audiotaped to make sure you are being rated correctly. The videotapes, will be erased within one year following your completion of the study. The videotapes will be used to help the investigators make sure that the counselors are following the correct procedures and may be used in future studies to help the investigators better understand the mood management and behavioral counseling treatments. No one but the study investigators or those delegated by the study investigators will be allowed to view the tapes and the identity of the participants will be kept strictly confidential. Staff that may be given permission by the study investigators to view the tapes include project staff, consultants that review and rate how well the study therapists giving the intervention follow study guidelines, and/or consultants that review how the assessments are given.

This is an investigational study. Up to 450 women will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Gestation: < or = 32 weeks pregnant at baseline
* Age: 16 years or older
* Smoking: at least a puff of a cigarette in the past 7 days & willing to set quit date that occurs before the end of treatment.
* English speaking & have a telephone
* Willing to attend all sessions and have no known complications that would adversely affect attendance
* Other: provide informed consent & agree to all assessments & study procedures

Exclusion Criteria:

* Current psychotherapy
* Involvement within one day of telephone screen with any smoking cessation activities other than those that are freely available in the public domain.
* History of/current medical condition, or any other factor, that, in the judgment of the Principal Investigator, would likely preclude completion of study requirements.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are pregnant smokers who may be under stress.
Sampling Method: Probability Sample
Enrollment: 338 (Actual)
Dates: Start 2004-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Prolonged Abstinence | 3 month assessments from end of treatment
  Prolonged abstinence assessed following treatment through 6 months postpartum to test effectiveness of health education versus a mood management treatment for helping pregnant women quit smoking.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Cinciripini, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org